CLINICAL TRIAL: NCT02452814
Title: Long-term Extension to a Phase 2, Open-Label, Clinical Trial of Miravirsen Sodium in Combination With Telaprevir and Ribavirin in Null Responders to Pegylated-Interferon Alpha Plus Ribavirin Subjects With Chronic Hepatitis C Virus Genotype 1 Infection
Brief Title: Long Term Extension Study is Designed to Monitor Long-Term Efficacy and Safety of Miravirsen Sodium in Combination With Telaprevir and Ribavirin in Subjects With Chronic Hepatitis C Virus Genotype 1 Infection
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: NP29710
Record Dates: First submitted 2015-05-11; First posted 2015-05-25 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: HCV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
Long Term Observational Extension Study Designed to Monitor Long-Term Efficacy and Safety of Miravirsen Sodium in Combination with Telaprevir and Ribavirin in Subjects with Chronic Hepatitis C Virus Genotype 1 Infection

ELIGIBILITY:
Inclusion Criteria:

- Participated in Study SPC3649-205 (this would include those who completed study SPC3649-205, those who discontinued or terminated the study early for whatever reason (including treatment failure) and those who opted to receive approved therapy for the treatment of HCV infection).

Exclusion Criteria:

* Those unwilling to provide informed consent for participation in this study.
* Subjects who have received investigational drug therapy after discontinuation, termination, or successful completion of Study SPC3649-205.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include null responder subjects with Chronic hepatitis C (CHC) genotype 1 virus infection who have participated in Study SPC3649-205.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with adverse changes in liver ultrasound results | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (2):
  - Methodist Transplant Physicians, Dallas, Texas
  - Research Specialists of Texas, Houston, Texas
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico